CLINICAL TRIAL: NCT00468559
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Treatment-withdrawal Study to Evaluate the Efficacy and Safety of Esomeprazole for the Treatment of Gastroesophageal Reflux (GERD) in Infants Aged 1 to 11 Months, Inclusive
Brief Title: Phase 3/Safety & Efficacy of Esomeprazole in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9614C00096
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-04

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: pediatrics; neonates
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Open Label Esomeprazole (Experimental): This is an open label, run-in phase. All patients received Esomeprazole.
  Interventions: Drug: Open Label Run In Esomeprazole
- Double Blind Esomeprazole (Experimental): This is the double blind withdrawal phase. Patients are randomized to active drug or placebo.
  Interventions: Drug: Double Blind Esomeprazole
- Double Blind Placebo (Placebo Comparator): This is the double blind withdrawal phase. Patients are randomized to active drug or placebo.
  Interventions: Drug: Double Blind Placebo

INTERVENTIONS:
Drug: Open Label Run In Esomeprazole — Esomeprazole magnesium in capsules dosing weight-dependent (2.5 mg - 10 mg)
  Arms: Open Label Esomeprazole
Drug: Double Blind Esomeprazole — Esomeprazole magnesium in capsules dosing weight-dependent (2.5 mg - 10 mg)
  Arms: Double Blind Esomeprazole
Drug: Double Blind Placebo — Double Blind Placebo
  Arms: Double Blind Placebo

SUMMARY:
The purpose of this study is to look at the improvement of a once a day dose of esomeprazole for reducing the signs and symptoms of infants with gastroesophageal reflux disease (GERD). This research study consists of a screening, open-label, and double-blind treatment withdrawal phase. The screening phase ensures the patient eligibility. No study medication is dispensed during the screening phase. During the open-label phase, patients are administered esomeprazole 2.5mg, 5.0mg or 10.0mg based on his/her weight. During the double-blind phase, the patients are administered either his/her open-label dose or placebo. Double-blind means neither the physician, parent, or patient will know if patient is taking esomeprazole or placebo. The patient will have an equal chance of receiving esomeprazole or placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients' parents must sign the informed consent prior to the beginning of any study-related procedures (according to local regulations)
* patients must have symptoms at study entry and have a clinical diagnosis of suspected GERD, symptomatic GERD, or GERD proven by a test called an endoscopy, a test using a long tube inserted in the body for diagnostic exams

Exclusion Criteria:

* patients who have used a PPI (proton pump inhibitors; used to reduce the amount of acid in the stomach) within 7 days before enrollment in the open label treatment phase (Day 0)
* patients with a history of acute life-threatening event

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ilueca, Study Director — AstraZeneca; Jennifer Heckman, Study Director — AstraZeneca; Jill McGuinn, Study Director — AstraZeneca
Locations (25):
- United States (14):
  - Research Site, Phoenix, Arizona
  - Research Site, Atlanta, Georgia
  - Research Site, Park Ridge, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Marrero, Louisiana
  - Research Site, Newton, Massachusetts
  - Research Site, Southfield, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Akron, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Chattanooga, Tennessee
  - Research Site, Roanoke, Virginia
- France (2):
  - Research Site, Lille
  - Research Site, Paris
- Germany (5):
  - Research Site, Bochum
  - Research Site, Greifswald
  - Research Site, Nurberg
  - Research Site, Potsdam
  - Research Site, Wuppertal
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Warsaw
  - Research Site, Wroclaw

REFERENCES:
- [Derived] Winter H, Gunasekaran T, Tolia V, Gottrand F, Barker PN, Illueca M. Esomeprazole for the Treatment of GERD in Infants Ages 1-11 Months. J Pediatr Gastroenterol Nutr. 2015 Jul;60 Suppl 1:S9-15. doi: 10.1097/MPG.0b013e3182496b35. PMID 26422097
- [Derived] Winter H, Gunasekaran T, Tolia V, Gottrand F, Barker PN, Illueca M. Esomeprazole for the Treatment of GERD in Infants Ages 1-11 Months. J Pediatr Gastroenterol Nutr. 2015 Jul;60 Suppl 1:S9-15. doi: 10.1097/MPG.0b013e3182496b35. PMID 26121349
- [Derived] Winter H, Gunasekaran T, Tolia V, Gottrand F, Barker PN, Illueca M. Esomeprazole for the treatment of GERD in infants ages 1-11 months. J Pediatr Gastroenterol Nutr. 2012 Jul;55(1):14-20. doi: 10.1097/MPG.0b013e3182496b35. PMID 22241513
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=440&filename=CSR-D9614C00096.pdf
- See also: CSR-D9614C00096.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=440&filename=CSR-D9614C00096.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged 1 to 11 months inclusive with a clinical diagnosis of suspected Gastroesophageal Reflux Disease (GERD), symptomatic GERD, or endoscopically proven GERD were enrolled across the USA France Germany and Poland. All patients were symptomatic at study entry.
Pre-assignment Details: All participants received 2-weeks open label esomeprazole (Open-label phase) according to baseline weight (3 to 5kg: 2.5mg; >5 to 7.5kg:5mg; >7.5-12kg:10mg). Following the open-label phase, those with symptom improvement of at least one category in the physician global assessment were eligible to be randomized into the withdrawal phase.
Groups:
- Open Label Esomeprazole: Open-label daily esomeprazole (2.5mg, 5mg or 10mg daily during open-label phase of the study, according to baseline weight). Eligible participants from the Open Label phase were randomized to the the double blind withdrawal phase.
Period: Open-label Treatment Phase
Arm/Group | Open Label Esomeprazole | Double Blind Esomeprazole | Double Blind Placebo
Started | 98 (All participants received open-label esomeprazole during this phase of the study) | 0 | 0
Completed | 80 (18 patients discontinued (were not randomized into the double-blind treatment withdrawal phase)) | 0 | 0
Not Completed | 18 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Lack of Efficacy | 9 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Period: Double-blind, Treatment-withdrawal Phase
Arm/Group | Open Label Esomeprazole | Double Blind Esomeprazole | Double Blind Placebo
Started | 0 | 39 | 41
Completed | 0 | 29 | 24
Not Completed | 0 | 10 | 17
Not completed — Lack of Efficacy | 0 | 8 | 17
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: Months] | 4.9 (2.6) | 4.9 (3.2) | 4.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 30 | 27 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Discontinuing Due to Symptom Worsening in the Randomized Treatment Withdrawal Phase (Treatment Withdrawal Phase Endpoint)
Description: Number of participants discontinuing during the 4-week of randomized double-blind withdrawal phase that met the pre-set definition of symptom worsening criteria.
Time Frame: Treatment-withdrawal phase (up to 4 weeks following randomization, or until earlier discontinuation from the study)
Population: reporting cumulative discontinuations
Measure: Number; unit: Participants
Groups:
- Double Blind Esomeprazole: In the double-blind treatment-withdrawal phase of the study, participants in this group received double-blind esomeprazole at the same dose they received in the preceeding open-label phase of the study.
- Double Blind Placebo: Participants in this group received placebo during the double-blind treatment withdrawal phase.
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 39 | 41
Participants
  Week 1 | 1 | 6
  Week 2 | 8 | 12
  Week 3 | 9 | 13
  Week 4 | 15 | 20

2. Secondary Outcome: Number of Participants Discontinuing Due to Any Reason, Including Symptom Worsening, in the Randomized Treatment Withdrawal Phase (Treatment Withdrawal Phase Endpoint)
Description: Number of participants discontinuing due to any reason was identical to the number of participants discontinuing due to symptom worsening (the primary assessment) when no participants discontinued due to reason other than symptom worsening.
Time Frame: Treatment withdrawal phase (up to 4 weeks following randomization, or until earlier discontinuation from the study)
Population: Reporting cumulative discontinuations. Results for the analysis of the secondary variable, time to discontinuation due to any cause, were identical to that found for the primary variable, time to discontinuation due to symptom.
Measure: Number; unit: Participants
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 39 | 41
Participants
  Week 1 | 1 | 6
  Week 2 | 8 | 12
  Week 3 | 9 | 13
  Week 4 | 15 | 20

3. Secondary Outcome: Treatment Successes at the End of the 4-week Double-blind Treatment Withdrawal Phase (Treatment Withdrawal Phase Endpoint).
Description: The number of participants reaching the end of the treatment withdrawal phase without discontinuing from the study (for any reason) or showing symptom worsening in the physician global assessment of Gastroesophageal Reflux Disease (GERD) symptoms. Based on the severity of symptoms reported by the parent/guardian in IVRS, the investigator provided the overall clinical impression of the patient's GERD-related symptoms over the last 7 days as:
  None Mild Moderate Severe
Time Frame: Treatment withdrawal phase (up to 4 weeks following randomization, or until earlier discontinuation from the study)
Measure: Number; unit: Participants
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 39 | 41
Participants | 24 | 21

4. Secondary Outcome: Physician's Global Assessment (PGA) of Gastroesophageal Reflux Disease (GERD) Symptoms (Treatment Withdrawal Phase Endpoint)
Description: Percentage of participants with Physician's Global Assessment (PGA) score at the final treatment withdrawal assessment in following categories: None (no symptoms), Mild, Moderate or Severe. The worst post-randomization Physician's Global Assessment (PGA) assessment during double blind phase is taken into account.
Time Frame: Treatment withdrawal phase (up to 4 weeks following randomization, or until earlier discontinuation from the study)
Measure: Number; unit: Percentage of participants
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 39 | 41
Percentage of participants
  None | 10.3 | 4.9
  Mild | 51.3 | 48.8
  Moderate | 25.6 | 31.7
  Severe | 12.8 | 14.6

5. Secondary Outcome: Severity of Vomiting/Regurgitation Symptoms as Reported by the Parent/Guardian (Treatment Withdrawal Phase Endpoint)
Description: Change from baseline in symptom severity (Severity is scored as 0-4 [none, mild moderate, severe]). For each participant, final severity score is the mean severity in the final 7-days, while baseline is the mean severity in the 7-day period up to and including randomization. Changes less than zero indicate improved severity versus baseline. Participants needed baseline measure and one additional post baseline measure to be included in analysis.
Time Frame: Treatment withdrawal phase (up to 4 weeks following randomization, or until earlier discontinuation from the study) Change was calculated from baseline to last measure obtained
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 37 | 40
Units on a scale | 0.040 (0.560) | 0.090 (0.610)

6. Secondary Outcome: Severity of Irritability Crying/Fussing Symptoms as Reported by the Parent/Guardian (Treatment Withdrawal Phase Endpoint)
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 37 | 40
Units on a scale | 0.060 (0.580) | 0.190 (0.590)

7. Secondary Outcome: Severity of Supraesophageal/Respiratory Disturbances (Coughing/Wheezing,Labored Breathing) as Reported by Parent/Guardian (Treatment Withdrawal Phase Endpoint)
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 37 | 40
Units on a scale | 0.120 (0.480) | 0.030 (0.580)

8. Secondary Outcome: Severity of Feeding Difficulties Reported by Parent/Guardian (Treatment Withdrawal Phase Endpoint)
Description: as for outcome 5
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Double Blind Esomeprazole | Double Blind Placebo
Number analyzed (Participants) | 37 | 40
Units on a scale | 0.090 (0.480) | 0.100 (0.610)

9. Secondary Outcome: Improvement in Physician's Global Assessment (PGA) Following Open-label Esomeprazole (Open-label Phase Endpoint)
Description: Number of patients who had an improvement of at least one category in the PGA at the end of open-label treatment with esomeprazole compared to baseline. Improvement in PGA was a pre-requisite for randomization into the randomized treatment withdrawal phase. Only patients with PGA at baseline and end of open-label are analyzed here.
Time Frame: Open-label treatment period (2 weeks)
Population: 95 patients received open-label esomeprazole during the open-label phase.
Measure: Number; unit: Participants
Groups:
- Open Label Esomeprazole: Open-label daily esomeprazole (2.5mg, 5mg or 10mg daily during open-label phase of the study, according to baseline weight)
Arm/Group | Open Label Esomeprazole
Number analyzed (Participants) | 95
Participants | 81

10. Secondary Outcome: Severity of Vomiting/Regurgitation Symptoms as Reported by the Parent/Guardian (Open-label Phase)
Description: Symptom severity (Severity is scored as 0-4 [none, mild moderate, severe]). For each participant, The score is the mean severity in each 7-day period.
Time Frame: Open Label phase (Screening plus two weeks)
Population: 84 patients were analyzed at the screening timepoint, 84 patients were analyzed at week 1 and 79 patients were analyzed at Week 2 due to discontinuations.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open Label Esomeprazole
Number analyzed (Participants) | 84
Units on a scale
  Screening | 1.42 (0.76)
  Week 1 | 1.14 (0.67)
  Week 2 | 1.00 (0.72)

11. Secondary Outcome: Severity of Irritability Crying/Fussing Symptoms as Reported by the Parent/Guardian (Open-label Phase Endpoint)
Description: as for outcome 10
Time Frame: Open Label Phase (Screening plus two weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open Label Esomeprazole
Number analyzed (Participants) | 84
Units on a scale
  Screening | 1.50 (0.67)
  Week 1 | 1.22 (0.68)
  Week 2 | 1.02 (0.74)

12. Secondary Outcome: Severity of Supraesophageal/Respiratory Disturbances (Coughing/Wheezing,Labored Breathing) as Reported by Parent/Guardian (Open-label Phase Endpoint)
Description: as for outcome 10
Time Frame: Open Label Phase (Screening plus two weeks)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open Label Esomeprazole
Number analyzed (Participants) | 84
Units on a scale
  Screening | 0.54 (0.69)
  Week 1 | 0.48 (0.61)
  Week 2 | 0.44 (0.69)

13. Secondary Outcome: Severity of Feeding Difficulties as Reported by Parent/Guardian (Open-label Phase Endpoint)
Description: as for outcome 10
Time Frame: Open Label Phase (Screening plus two weeks)
Population: 83 patients were analyzed at the screening timepoint, 83 patients were analyzed at week 1 and 78 patients were analyzed at Week 2 due to discontinuations.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open Label Esomeprazole
Number analyzed (Participants) | 83
Units on a scale
  Screening | 1.16 (0.76)
  Week 1 | 0.94 (0.71)
  Week 2 | 0.83 (0.76)

ADVERSE EVENTS:
Groups:
- Open-label Phase: Open-label daily esomeprazole (2.5mg, 5mg or 10mg daily during open-label phase of the study, according to baseline weight).
- Double Blind Esomeprazole; Double Blind Placebo: Eligible participants from the Open Label phase were randomized to the the double blind withdrawal phase.
Arm/Group | Open-label Phase | Double Blind Esomeprazole | Double Blind Placebo
Serious Adverse Events (participants affected / at risk) | 4/98 | 3/39 | 0/41
Other Adverse Events (participants affected / at risk) | 26/98 | 19/39 | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Phase (N=98) | Double Blind Esomeprazole (N=39) | Double Blind Placebo (N=41)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chlamydial Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Poor Peripheral Circulation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rotavirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Phase (N=98) | Double Blind Esomeprazole (N=39) | Double Blind Placebo (N=41)
Bronchitis (Infections and infestations) | 4 | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 2
Flatulence (Gastrointestinal disorders) | 1 | 2 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3
Otitis Media (Infections and infestations) | 2 | 2 | 1
Pyrexia (General disorders) | 4 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rhinitis (Infections and infestations) | 3 | 4 | 3
Teething (Gastrointestinal disorders) | 4 | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 6 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2
Ear Infection (Infections and infestations) | 0 | 2 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less